CLINICAL TRIAL: NCT04163601
Title: NTM-net Study: Liposomal Amikacin Inhalation in M.Abscessus Patients
Brief Title: Liposomal Amikacin Inhalation in M.Abscessus Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: European network (http://www.ntm-net.org/index.php/ntm-net) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0487
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2019-11

CONDITIONS: M.Abscessus Pulmonary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mycobacterium abscessus is one of the many species of non-tuberculous mycobacteria. M. abscessus infections are known to be common in patients with cystic fibrosis (CF). Mycobacterium abscessus yields poor cure rates. Liposomal amikacin inhalation (LAI) might be a good alternative for intravenous treatment as the first results with mycobacterium avium treatment yield good results.

The objective of this study is to summarize the clinical data of patients with M.abscessus treated with LAI on compassionate use basis to assess treatment outcomes

ELIGIBILITY:
Inclusion criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* ATS diagnostic criteria for M.abscessus pulmonary disease
* > 12 years
* Patients with CF/COPD or other underlying disease
* LAI use for more than 3 weeks

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

• Extra-pulmonary or disseminated disease

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with M. abscessus disease
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-11-30 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
culture conversion | 1 day
  Main study endpoints will consist of microbiological cure, clinical cure and treatment culture conversion at the end of treatment. Treatment outcome definitions according to the NTM net consensus are used

SECONDARY OUTCOMES:
clinical cure | 1 day
  Main study endpoints will consist of microbiological cure, clinical cure and treatment culture conversion at the end of treatment. Treatment outcome definitions according to the NTM net consensus are used

CONTACTS AND LOCATIONS:
Overall Officials: Raphael CHIRON, PU-PH, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC